CLINICAL TRIAL: NCT03964883
Title: Infliximab Blood Test in Crohn's Disease
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: LAP CROHN INFLIXIMAB
Record Dates: First submitted 2019-05-22; First posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ano-perineal lesions are the first signs of Crohn's disease in 1/3 to 1/2 of cases. They are most often associated with a poor prognosis of the disease and their management is complex and difficult because of the dilapidated and recurrent nature of lesions with significant repercussions on continence and quality of life.

The treatment of these lesions is most often medical and surgical, consisting of drainage of the suppurative lesions and/or the use of biotherapy +/- combined with an immunosuppressant.

DETAILED DESCRIPTION:
Pharmacological dosages of biotherapies show a significant correlation between the highest rates and the achievement of clinical and endoscopic remission. Therapeutic monitoring by dosing the residual levels of these biotherapies and specific antibodies, particularly in the event of loss of response in order to adapt the treatment, has become common for luminal damage. Among these biotherapies, infliximab is the first-line treatment, particularly for ano-perineal disease. Effective therapeutic levels are known for luminal damage and must be between 3 and 7 mcg/ml but these levels have not yet been determined for ano-perineal damage. There are only two recently published studies available that suggest levels probably significantly higher than those required for luminal damage ≥ 10 mcg/l

ELIGIBILITY:
Inclusion Criteria:

* All patients followed for Chron's diseases within Groupe Hospitalier Paris Saint-Joseph (GHPSJ) and treated with Infliximab for at least 6 months.

Exclusion Criteria:

* All patients with therapeutic compliance problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed for Crohn's disease and treated with Infliximab
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Identify doses and residual levels of infliximab in patients affected by ano-perineal Crohn's disease in remission | Time of inclusion
  doses and residual levels of infliximab in remission patients will be collected to determine minimum, maximum and average values.

SECONDARY OUTCOMES:
Compare doses and residual rates of infliximab in patients affected by Crohn's disease in remission with luminal impairment alone versus ano-perineal +/- luminal | Time of inclusion
  Doses and infliximab's residual levels will be collected from patients affected by Crohn's disease in remission with luminal alone and from patients in remission with ano-perineal +/- luminal for comparison
Evaluate the proportion of patients in luminal remission with active ano-perineal disease | Time of inclusion
  Calculation of patient's proportion with active ano-perineal disease on total of all patients in luminal remission.
Compare residual doses and infliximab levels in patients with ano-perineal disease in remission versus active | Time of inclusion
  Infliximab doses, infliximab residual levels will be collected from patients affected by Crohn's disease with ano-perineal involvement to compare remission patients and patients with active disease.
Anti-infliximab antibodies presence (yes/no) in patients with ano-perineal disease in remission versus active | Time of inclusion
  Anti-infliximab antibodies will be collected from patients affected by Crohn's disease with ano-perineal involvement to compare remission patients and patients with active disease.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Fathallah, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, France

REFERENCES:
- [Result] Davidov Y, Ungar B, Bar-Yoseph H, Carter D, Haj-Natour O, Yavzori M, Chowers Y, Eliakim R, Ben-Horin S, Kopylov U. Association of Induction Infliximab Levels With Clinical Response in Perianal Crohn's Disease. J Crohns Colitis. 2017 May 1;11(5):549-555. doi: 10.1093/ecco-jcc/jjw182. PMID 28453755
- [Result] Yarur AJ, Kanagala V, Stein DJ, Czul F, Quintero MA, Agrawal D, Patel A, Best K, Fox C, Idstein K, Abreu MT. Higher infliximab trough levels are associated with perianal fistula healing in patients with Crohn's disease. Aliment Pharmacol Ther. 2017 Apr;45(7):933-940. doi: 10.1111/apt.13970. Epub 2017 Feb 17. PMID 28211593
- [Result] Mitrev N, Kariyawasam V, Leong RW. Editorial: infliximab trough cut-off for perianal Crohn's disease - another piece of the therapeutic drug monitoring-guided infliximab dosing puzzle. Aliment Pharmacol Ther. 2017 May;45(9):1279-1280. doi: 10.1111/apt.14020. No abstract available. PMID 28370040